CLINICAL TRIAL: NCT00260988
Title: Tinzaparin Versus Dalteparin for Perioperative Thromboembolic Prophylaxis in Patients With Dialysis Dependent Renal Disease- A Canadian Multicentre Trial
Brief Title: A Comparison of Dalteparin and Tinzaparin for Prevention of Blood Clots in Hemodialysis Patients on Oral Anticoagulants Having Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2003391-01H
Record Dates: First submitted 2005-11-30; First posted 2005-12-02 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2009-07

CONDITIONS: Thromboembolism; Hemodialysis
Keywords: Prophylaxis; Thromboembolic disease; End stage renal disease; Hemodialysis; Pharmacokinetics; Low Molecular Weight Heparin; Innohep; Tinzaparin; Fragmin; Dalteparin; Anti Xa; INR; Oral anticoagulation; warfarin; Coumadin
MeSH Terms: conditions — Thromboembolism; Kidney Failure, Chronic | interventions — Dalteparin; Tinzaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dalteparin (Active Comparator): Dalteparin 200 IU/kg/day for three days prior to surgery and dalteparin 5000IU daily for 3-5 days post-surgery
  Interventions: Drug: Fragmin (dalteparin)
- Tinzaparin (Active Comparator): Tinzaparin 175 IU/kg/day for three days prior to surgery and Tinzaparin 4500 IU for 3-5 days post surgery
  Interventions: Drug: Innohep (tinzaparin)

INTERVENTIONS:
Drug: Fragmin (dalteparin) — 200 IU/Kg/Day administered subcutaneously for three days prior to but not including the day of the surgery
  Arms: Dalteparin
Drug: Innohep (tinzaparin) — 175 IU/kg/Day administered subcutaneously for three days prior to but not including the day of the surgery
  Arms: Tinzaparin

SUMMARY:
The purpose of this study is to better understand if either dalteparin or tinzaparin is a better drug to use in dialysis patients on blood thinners who are at high risk of developing blood clots and need surgery.

DETAILED DESCRIPTION:
A prospective multicenter randomised trial involving 60 consecutive eligible and consenting patients from teaching hospitals in Canada. Patients will be randomised to either tinzaparin or dalteparin to investigate the pharmacokinetics of both low molecular weight heparins (LMWH) perioperatively in a special population, namely end stage renal disease (ESRD) dialysis patients.

To date although there exists evidence to suggest tinzaparin may be safe in patients on hemodialysis, LMWHs as a group have not been investigated in the perioperative setting in these patients. This protocol has been developed so that the pharmacokinetic behaviour of tinzaparin and dalteparin can be compared but also so that the duration off warfarin is minimised. Therapeutic doses of LMWH are administered pre-procedure during as much time of the period as possible that oral anticoagulation is sub-therapeutic.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Patients aged >= 18 with end stage renal disease requiring chronic hemodialysis (HD) three times a week and clinically stable on HD for 4 weeks (x 4 wks)
* Patients requiring active oral anticoagulation for prosthetic heart valves, recent deep vein thrombosis >= 1 month, or patients with atrial fibrillation and a major risk factor (previous transient ischemic attack [TIA] or stroke, high blood pressure, diabetes, aged >= 75, moderate/severe left ventricle dysfunction) who require elective non-cardiac surgery or an invasive procedure with reversal of their anticoagulant therapy.

Exclusion Criteria:

* Evidence of active bleeding prior to stopping warfarin
* Hemoglobin <= 90 or platelet count <= 100x10^9/L
* Uncontrolled hypertension or stroke within 6 months of study commencement
* Spinal or neurosurgery
* Eye surgery (excluding cataract surgery)
* Life expectancy less than 3 months
* Patients requiring cardiac surgery
* Presence of active duodenal ulcer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2003-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Primary outcome will be the comparison of the pharmacokinetic profiles of dalteparin and tinzaparin in patients on hemodialysis in the setting of perioperative anticoagulation for thromboembolic prophylaxis. Specifically pre-dialysis anti-Xa levels post | Pre-dialysis following the third dose of LMWH
  Anti-Xa levels were drawn pre-dialysis (at a timepoint that was within 20-24hrs post- LMWH dose) and post- dialysis

SECONDARY OUTCOMES:
The frequency of surgery cancellation | Cumulatively collected at end of study
  We will collect data on reasons why surgeries were cancelled in this patient population
Bleeding complications | Any reported and elicited bleeding event will be captured throughout the study period

CONTACTS AND LOCATIONS:
Overall Officials: Marc Rodger, MD, MSc, Principal Investigator — OHRI
Locations (2):
- Canada (2):
  - St. Joseph's Healthcare, Hamilton, Ontario
  - The Ottawa Hospital, Ottawa, Ontario

REFERENCES:
- [Derived] Natale P, Palmer SC, Ruospo M, Longmuir H, Dodds B, Prasad R, Batt TJ, Jose MD, Strippoli GF. Anticoagulation for people receiving long-term haemodialysis. Cochrane Database Syst Rev. 2024 Jan 8;1(1):CD011858. doi: 10.1002/14651858.CD011858.pub2. PMID 38189593